CLINICAL TRIAL: NCT05742594
Title: A Phase 1, Open-label, Randomized, 4-Way Crossover Pivotal Study to Assess the Bioequivalence of Four Different Oral Tablet Formulations of Lazertinib (JNJ-73841937) in Healthy Adult Participants
Brief Title: A Study of Four Different Oral Tablet Formulations of Lazertinib (JNJ-73841937) in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CR109315; 73841937NSC1009 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2023-02-15; First posted 2023-02-24 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-06

CONDITIONS: Healthy
MeSH Terms: interventions — lazertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Intervention Sequence: ADBC (Experimental): Participants will receive intervention A (lazertinib reference formulation) on Day 1 of intervention Period 1, followed by intervention D (lazertinib test formulation) on Day 1 of intervention Period 2, followed by intervention B (lazertinib test formulation) on Day 1 of intervention Period 3 followed by intervention C (lazertinib test formulation) on Day 1 of Intervention Period 4. There will be a wash-out period of at least 14 days and up to 21 days between each intervention period.
  Interventions: Drug: Lazertinib
- Intervention Sequence: BACD (Experimental): Participants will receive intervention B (lazertinib test formulation) on Day 1 of intervention Period 1, followed by intervention A (lazertinib reference formulation) on Day 1 of intervention Period 2, followed by intervention C (lazertinib test formulation) on Day 1 of intervention Period 3 followed by intervention D (lazertinib test formulation) on Day 1 of intervention Period 4. There will be a wash-out period of at least 14 days and up to 21 days between each intervention period.
  Interventions: Drug: Lazertinib
- Intervention Sequence: CBDA (Experimental): Participants will receive intervention C (lazertinib test formulation) on Day 1 of intervention Period 1, followed by intervention B (lazertinib test formulation) on Day 1 of intervention Period 2, followed by intervention D (lazertinib test formulation) on Day 1 of intervention Period 3 followed by intervention A (lazertinib reference formulation) on Day 1 of intervention Period 4. There will be a wash-out period of at least 14 days and up to 21 days between each intervention period.
  Interventions: Drug: Lazertinib
- Intervention Sequence: DCAB (Experimental): Participants will receive intervention D (lazertinib test formulation) on Day 1 of intervention Period 1, followed by intervention C (lazertinib test formulation) on Day 1 of intervention Period 2, followed by intervention A (lazertinib reference formulation) on Day 1 of intervention Period 3 followed by intervention B (lazertinib test formulation) on Day 1 of intervention Period 4. There will be a wash-out period of at least 14 days and up to 21 days between each intervention period.
  Interventions: Drug: Lazertinib

INTERVENTIONS:
Drug: Lazertinib — Lazertinib will be administered orally.
  Other Names: JNJ-73841937

SUMMARY:
The purpose of this study is to assess the bioequivalence of four different lazertinib oral tablet formulations in healthy adult participants under fasted condition.

ELIGIBILITY:
Inclusion Criteria:

* Healthy on the basis of physical examination, medical history (at screening only), vital signs, and 12-lead electrocardiogram (ECG) performed at screening and at admission to the study site
* All female participants must have a negative highly sensitive serum Beta-human chorionic gonadotropin (Beta-HCG) at screening and on Day -1 of Intervention Period 1
* A male participant must agree not to donate sperm for the purpose of reproduction during the study and for a minimum of 6 months after receiving the last dose of study intervention
* Must sign an informed consent form (ICF) indicating that the participant understands the purpose of, and procedures required for, the study and is willing to participate in the study
* Female participants must be postmenopausal or surgically sterile

Exclusion Criteria:

* History of stomach or intestinal surgery or resection, including cholecystectomy, that would potentially alter absorption or excretion of orally administered drugs
* History of malignancy within 5 years before screening
* Known allergies, hypersensitivity, or intolerance to lazertinib or its excipients
* Participant has a history of clinically significant allergies
* Had major surgery, (for example, requiring general anesthesia) within 8 weeks before screening, or will not have fully recovered from the surgery, or has surgery planned during the time the participant is expected to participate in the study or within 4 weeks after the last dose of study intervention administration

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2023-01-03 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-04-03 (Actual)

PRIMARY OUTCOMES:
Interventions A, B and C: Maximum Observed Plasma Concentration (Cmax) of Lazertinib | Pre dose up to 168 hours post dose
  Cmax is defined as maximum observed plasma concentration.
Interventions A, B and C: Area Under the Plasma Concentration-time Curve from Time 0 to 72 Hours (h) (AUC[0-72h]) of Lazertinib | Pre dose up to 168 hours post dose
  AUC (0-72h) is the area under the plasma concentration-time curve from time 0 to 72 hours.

SECONDARY OUTCOMES:
Interventions A and D: Maximum Observed Plasma Concentration (Cmax) of Lazertinib | Pre dose up to 168 hours post dose
  Cmax is defined as maximum observed plasma concentration.
Interventions A and D: Area Under the Plasma Concentration-time Curve from Time of 0 to 72 Hours [AUC (0-72h)] of Lazertinib | Pre dose up to 168 hours post dose
  AUC (0-72h) is the area under the plasma concentration-time curve from time 0 to 72 hours.
Number of Participants With Adverse Events (AEs) | Up to 14 weeks
  AE is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.
Number of Participants With Serious Adverse Events (SAEs) | Up to 14 weeks
  A SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Number of Participants With AEs by Severity | Up to 14 weeks
  Number of participants with AEs by severity will be reported. Severity will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0. Severity scale ranges from grade 1 (mild) to grade 5 (death). Grade 1= mild, Grade 2= moderate, Grade 3= severe, Grade 4= life-threatening and Grade 5= death related to adverse event.
Number of Participants With Change From Baseline in Clinical Laboratory Test Values | Up to 14 weeks
  Number of participants with change from baseline in clinical laboratory test values (including hematology and clinical chemistry) will be reported.
Number of Participants With Change From Baseline in 12-lead Electrocardiograms (ECGs) | Up to 14 weeks
  Number of participants with change from baseline in 12-lead ECGs will be reported.
Number of Participants With Change From Baseline in Vital Signs | Up to 14 weeks
  Number of participants with change from baselines in vital signs (including temperature [oral], pulse/heart rate, respiratory rate, and blood pressure) will be reported.
Number of Participants With Change From Baseline in Physical Examination | Up to 14 weeks
  Number of participants with change from baseline in physical examination (including height and body weight) will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trail, Study Director — Janssen Research & Development, LLC
Locations (1):
- Celerion, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency